CLINICAL TRIAL: NCT00148434
Title: A Pilot Randomised Controlled Trial to Assess the Impact on Blood Pressure Control of Empowering Patients to Become Involved in Their Own Blood Pressure Management.
Brief Title: Study on Impact of Patient-Held Guidelines on Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ashgrove Research Practice (Other)
Collaborators: University of Edinburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OOB/3/19/F25; OOB/3/19/F25 CSO
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: hypertension; guidelines; patient empowerment; anxiety
MeSH Terms: conditions — Hypertension; Patient Participation; Anxiety Disorders

INTERVENTIONS:
Behavioral: Patient-held guideline for hypertension

SUMMARY:
While patient held guidelines for the management of chronic diseases have been employed in some countries. There is little evidence of their effectiveness in improving patient outcomes. We hypothesised that a patient held guideline on the management of hypertension combined with a specific exhortation to patients to challenge their medical care where the guidelines did not appear to have been applied would improve blood pressure control, lower average blood pressure, lower average cholesterol, increase the appropriate use of statins and aspirin, and have no impact on patient anxiety. Patients were randomised to the guideline or to standard hypertension information. Measures of anxiety were taken at baseline 2 weeks and one year, blood pressure and cholesterol was measured at one year and case notes examined to determine appropriate statin and aspirin usage.

DETAILED DESCRIPTION:
Prevention and treatment of hypertension and target organ disease remain important public health challenges which must be addressed (SIGN 2001). There is sound evidence that control of hypertension can significantly reduce the incidence of stroke and cardiac events (Mulrow and Pignone 2001). National guidelines for the identification and treatment of hypertension have been issued (Ramsey et al 1999, SIGN 2001) and a local version of the national guidelines has been issued to all GPs in Lothian. However, although there is evidence that most patients with hypertension are identified, many do not have their hypertension adequately controlled (Colhoun et al 1998), and GPs are reluctant to treat mild hypertension or hypertension in the elderly (Dickerson et al 1995a,b, Frijlen et al 2001).

Without additional interventions to encourage change in medical practice, the effects of clinical guidelines are generally limited (Effective Health Care 1994, Oxman et al 1995). A large number of additional interventions have been used to encourage the adoption of clinical guidelines including continuing medical education, dissemination of educational materials, educational outreach, local opinion leaders, audit and feedback, manual or computerised reminders, mass media campaigns, continuous quality improvement programmes (Effective Health Care 1999). All have some effect, but none are overwhelmingly successful or effective in all circumstances (Effective Health Care 1999, Davies et al 1995, Grimshaw et al 1995) It is suggested that multiple interventions may be more effective than single ones (Wensing and Grol 1994, Greco and Eisenberg 1993).

There is increasing evidence that in Primary Care patients' expectations have a significant effect on the treatment they get from their GP (Tomlin et al 1999, Howitt and Armstrong 1999). Mass media campaigns targeting patients have been found to influence professional practice (Grilli et al 2000). However, evaluation of the effect of locally provided patient information has been limited to the effect that it has on patient behaviour (e.g. compliance with dietary advice or medication) and not on the effect in may have on medical practice.

One initiative, which has not been fully evaluated, is distribution of the guidelines to patients. The large AHCPR guideline programme in the United States included the full guideline, a summary for professionals and a summary for patients (Colling 1994). Evaluation appeared to be limited to the distribution of these guidelines and the impact on practice was not measured (Colling 1994). When the Scottish (SIGN) clinical guideline programme was initiated much of the AHCPR methodology was adopted and acknowledged, but the patient guideline was not included. The purpose of this study is to evaluate the effect of providing patients with a clinical guideline (edited to be understandable to a lay person) on the overall management and control of their hypertension coupled with an explicit exhortation from the medical team to become involved in their own care.

3. Trial objectives and purpose: The trial aims to determine if the provision of a patient guideline on the management of hypertension.

1. Improves control of hypertension
2. Improves compliance by doctors with established guidelines
3. Increases patient anxiety

Three research questions have been set up in an attempt to meet these aims. Does provision of a patient guideline on the management of hypertension along with explicit exhortation to patients to challenge care that does not meet the guideline.

1. Improve control of hypertension, as evidence by average blood pressure achieved and numbers of patients who achieve control (i.e. BP < 150/90)
2. Improve compliance by doctors with established guidelines as evidenced by recorded calculation of 10 year cardiovascular risk, appropriate use of aspirin and cholesterol lowering agents, checking of cholesterol and level of blood cholesterol achieved, appropriate checking of urea and electrolytes and frequency of blood pressure monitoring.
3. Increase patient anxiety.

   4. Trial design:

a) A randomised trial has been set up to assess these research questions.

5. Selection and withdrawal of subjects:

a) All hypertensive patients from the Ashgrove Health Centre Blood Pressure Clinic (435) for whom recent baseline information on their blood pressure and control is available (these data were recently collected for an extensive audit) will be selected for invitation to take part in the study. All will be sent an invitation/ information letter to their home address asking them to consent to the study Those participants who consent to the study will also be asked to complete a questionnaire to measure anxiety (Hospital Anxiety and Depression Scale: HADS) and return it to the surgery using an SAE. Those who fail to return a response will be sent a reminder in two weeks. Information booklets will be sent to all participants who have consented (whether their anxiety questionnaire has been returned or not).

6. Treatment of subjects:

a) All hypertensive patients( at least one systolic BP > 150) in Ashgrove Health Centre for whom recent baseline information is available will be invited to take part in this study. As there are many households (approx. 30) with more than one hypertensive patient, randomisation will take place at household, rather than individual level, so that people living at the same address will receive the same treatment. Participants will be randomised into two groups (using a random number generator). One group will receive a detailed guideline and record card derived from the Lothian Hypertension Guideline which gives general information about blood pressure, but also provides the patient with clear guidelines as to how their blood pressure should be managed by medical and nursing staff and a clear exhortation to question their care if the guideline is not being adhered to (see attached draft). They will also be given a standard, high quality patient information booklet produced by the British Hypertension Society. The second group will be given the British Hypertension Society booklet only . This group will not be specifically exhorted to challenge their care in the same way as the other group.

Doctors in the study will not be told to treat the groups differently. We anticipate a Hawthorn effect in that doctors will inevitably be sensitised to comply with guidelines more rigorously for both groups.

All patients will be sent a letter explaining the study, a consent form and a Hospital Anxiety and Depression Score questionnaire. Those wishing to take part in the study will be asked to return the consent form and questionnaire in the accompanying stamped addressed envelope.

Patients will then be sent the booklet and in the intervention groups case the booklet and guideline. A further HADS score will be sent two weeks after the guideline to identify any immediate anxiety caused by the guideline.

All patients will be called in at the end of a year for BP measurement. Case notes will be searched for records of BP monitoring, cardiovascular risk recording, cholesterol estimation, appropriate use of cholesterol lowering agents, appropriate use of aspirin, actual blood cholesterol level, appropriate checking of Urea and Electrolytes. Patients will be asked to complete a further HADS and a questionnaire which ask them how they found the intervention and their perception of their involvement in the management of their blood pressure. Doctors and nurses in the practice will be interviewed about their experience in relation to the project in terms of perceived increased workload and their experience (if so perceived) of managing consultations with empowered patients.

7. Statistics:

a) This project is a pilot and will help in calculating the power of future studies. However, we have calculated that this study has 80% power to detect as significant at the 5% level differences in mean blood pressure of the order of 2-3 mm Hg, or of 10-15% in the percentage of patients achieving BP targets. Statistical analyses will be carried out by Dr. Rob Elton, statistical consultant.

8. Data handling and record keeping:

1. All patient records will be pulled and perused only by the research nurse who is a member of staff at Ashgrove Health Centre. While research data are being collected, they will be kept completely confidential and stored on a password protected computer at Ashgrove Health Centre. Once all data are collected, they will be anonymised. No patients will be identifiable from any of the results, published or otherwise.
2. Audio taping of focus groups with staff on completion of the study will take place. The tapes will be kept in a locked filing cabinet in the Department of General Practice at the University of Edinburgh. On completion of tape transcription, the tapes will be destroyed. All transcripts of tapes will be anonymised so that staff participants will not be identifiable.

Colhoun et al (1998) Blood pressure screening, management and control in England: results from the health survey for England 1994. J Hypertens 16(6):747-52

Colling 1994). Colling J (1994). An update on the AHCPR guideline implementation. Nurs Pract Forum,5,134-137

Davis DA Taylor-Vaisey MLS (1997) Translating guidelines into practice. Can Med Assoc J 157, (4) 408-416

Dickerson JE, Brown MJ (1995a). Influence of age on general practitioners' definition and treatment of hypertension. BMJ, 310, 574

Dickerson JE, Garratt CJ, Brown MJ (1995b) Management of hypertension in general practice: agreements with and variations from the British Hypertension Society guidelines. J Hum Hypertens; 9: 835-9

Effective health Care (1994) No 8 - Implementing Clinical Practice Guidelines. Leeds: University of Leeds

Effective Health Care (1999) 5 (1) Getting evidence into practice. York: NHS Centre for Reviews and Dissemination

Frijlen B, Spes T, Lobo C, Hulscher E et al. (2001) Blood pressure control in treated hypertensive patients: clinical performance of General Practitioners. BJGP 51(462), 9-15

Greco PJ, Eisenberg JM (1993) Changing physician's practices. New England Journal of Medicine, 329 (17), 1271-1274

Grilli R, Freemantle N, Minozzi S, Domenighetti G, Finer D.(2001) Mass media interventions: effects on health services utilisation (Cochrane Review). In: The Cochrane Library, Issue 2, . Oxford: Update Software.

Grimshaw J, Freemantle N, Wallace S, Russell I, Hurwitz B, Watt I, Long A, Sheldon T (1995) Developing and implementing clinical guidelines. Quality in Health Care, 4 55-64

Heaney, D., Wyke, S., Wilson, P., Elton, R. and Rutledge, P. (2001) Assessment of impact of information booklets on use of healthcare services: randomised control trial. British Medical Journal 322, 1-5.

Howitt A, Armstrong D (1999) Implementing evidence based medicine in general practice: audit and qualitative study of antithrombotic treatment for atrial fibrillation. BMJ, 318, 1324-1327

Mulrow CD, Pignone M (2001) What are the elements of good treatment for hypertension? BMJ, 322,1107-9

Oxman AD, Thomson MA, Davis DA, et al (1995) No magic bullets: a systematic review of 102 trials of interventions to improve professional practice. CMAJ, 153,1423-31

Ramsey LE, Williams B, Johnston GD et al (1999). British Hypertension Society guidelines for the management of hypertension: report of the third working party of the British Hypertension Society. J Hum Hypertens; 13:569-92

SIGN (2001) Hypertension in older people. Edinburgh: SIGN

Tomlin Z, Humphrey C, Rogers S (1999) General practitioners perceptions of effective health care. Brit Med J, 318, 1532-5

Wensing M. Grol R (1994) Single and combined strategies for implementing changes in primary care: a literature review. Quality in Health Care 6 (2) 115-132

Wilkie, T. (2001) Commentary: Public opinion may force researchers to seek "opt-in" consent for all studies. British Medical Journal 322, 5.

ELIGIBILITY:
Inclusion Criteria:

* All patients on the hypertension register of the practice

Exclusion Criteria:

* Patients unable to consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2002-01; Study Completion 2003-03

PRIMARY OUTCOMES:
Proportion of patients with systolic blood pressure <150 and diastolic blood pressure <90

SECONDARY OUTCOMES:
Average systolic blood pressure
Average cholesterol
Proportion of patients with cholesterol < 5.0mmol/l
Hospital Anxiety and Depression Score
Proportion with appropriate use of aspirin and statins according to UK guideline
Satisfaction with care
Perception of involvement with decision making

CONTACTS AND LOCATIONS:
Overall Officials: Brian McKinstry, MD, Principal Investigator — University of Edinburgh
Locations (1):
- Ashgrove Health Centre, Blackburn West Lothian, United Kingdom